CLINICAL TRIAL: NCT00556907
Title: Targeted Intra-Operative Radiotherapy for the Management of Ductal Carcinoma In-Situ of the Breast (TARGIT-DCIS Trial): Use of Mammography and Breast MRI to Identify Candidates for IORT.
Brief Title: Targeted Intra-Operative Radiotherapy for the Management of Ductal Carcinoma In-Situ of the Breast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-06-9
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: DCIS; To evaluate Preoperative mammagraphy and MRI to select candiates with DCIS for IORT
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 1 (Other): Patients will receive IORT
  Interventions: Radiation: Intraoperative radiotherapy; Device: Intraoperative radiotherapy

INTERVENTIONS:
Radiation: Intraoperative radiotherapy — 20Gy to surface of tumor bed and 5Gy at depth of 1cm from surface of tumor bed
  Other Names: Intrabeam Photon Radiosurgery System and Applicators
Device: Intraoperative radiotherapy — 20gy to tumor bed, 5gy at depth of 1cm from surface of tumor bed
  Other Names: Intrabeam Photon Radiosurgery

SUMMARY:
We hypothesize that the combination of mammography and CE-MRI will improve the surgeon and radiologist's ability to define extent of disease prior to surgical resection, improve the odds of obtaining clear surgical margins, and increase the efficacy of IORT delivered immediately after initial surgical resection. In this investigation, we will determine whether or not patients deemed eligible for 'immediate" IORT based on mammography and CE-MRI can be successfully treated without the need for re-excision or additional radiotherapy due to inadequate surgical margins.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven DCIS, mammographic and CE-MRI evidence of DCIS measuring great then equal to 4cm, and a desire to receive breast conserving therapy, will be considered for participation in this study.
* Patient history, physical examination findings, and demographics (sex, age, height, weight, bra size, etc.) will be performed and documented.

Inclusion Criteria for Initial Registration (all patients cohorts):

All cohorts

* Signed informed consent and HIPAA documents
* Female sex
* Age great then equal to 40 years
* Localized ductal carcinoma in situ
* Clinically and/or histologically negative axillary lymph nodes
* No imaging or clinical findings suggestive of invasive carcinoma.

Cohort 1 (Immediate IORT group)

* Localized DCIS measuring less then equal to 4 cm on preoperative imaging.
* Cohort 2 (Delayed IORT group)
* Localized DCIS measuring less then equal to4 cm or less on surgical pathology
* Delayed IORT could be performed for the explicit purpose of administering IORT or performed following re-excision of a previously operated breast to achieve clear surgical margins.
* This cohort includes patients who were excluded from immediate IORT based on pre-operative imaging suggesting ineligibility for immediate IORT, but who are subsequently found to meet histological criteria (localized DCIS less then equal to 4 cm and no invasive cancer) for IORT based on surgical pathology.
* Unifocal microinvasive (T1mic or invasive focus less then equal to 1mm in maximal diameter) is allowed following initial WLE if surgical pathology margins were less then equal to2 mm for both the invasive and non-invasive components.
* Delayed IORT must be performed within 3 months of initial WLE.
* Cohort 3 Subjects who received IORT at the time of initial WLE but whose surgical pathology showed them to be unsuitable candidates for IORT alone on the basis of:
* DCIS measuring greater than 5 cm on surgical pathology.
* T1a (less than 1 mm) or larger invasive carcinoma associated with extensive DCIS.
* Surgical margins width less than1 mm.

Exclusion Criteria:

* Male sex
* Age less than 40
* DCIS associated with any evidence of microinvasion or invasive carcinoma on pre-operative imaging or core biopsy of the breast or axillary nodes.
* DCIS that is multicentric in the ipsilateral breast. Multicentricity will be defined at 2 or more lesions separated by more than 3 cm in the same breast.
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* DCIS associated with diffuse suspicious or indeterminate microcalcifications
* Pregnancy or lactation
* Collagen vascular diseases, including Systemic lupus erythematosus, Systemic sclerosis (scleroderma), CREST Syndrome (calcinosis, Raynaud phenomenon, esophageal dysfunction, sclerodactyly, telangiectasia, and the presence of anticentromere antibodies), polymyositis, dermatomyositis with a CPK level above normal or with an active skin rash, inclusion-body myositis, or amyloidosis
* Serious psychiatric or addictive disorders

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Macdonald, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Hickey BE, Lehman M. Partial breast irradiation versus whole breast radiotherapy for early breast cancer. Cochrane Database Syst Rev. 2021 Aug 30;8(8):CD007077. doi: 10.1002/14651858.CD007077.pub4. PMID 34459500

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraoperative Radiotherapy: Patients will receive IORT
  Intraoperative radiotherapy: 20Gy to surface of tumor bed and 5Gy at depth of 1cm from surface of tumor bed
  Intraoperative radiotherapy: 20gy to tumor bed, 5gy at depth of 1cm from surface of tumor bed
Period: Overall Study
Arm/Group | Intraoperative Radiotherapy
Started | 36
Completed | 35
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Radiotherapy
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: Years] | 57 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Reoperation (Re-excision or Mastectomy) Rates Following WLE or IORT
Description: These are the rates of reoperation for re-excision or mastectomy following Wide Local Excision (WLE) or Intraoperative Radiation Therapy (IORT). The number of patients who required reoperation were reported below.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Radiotherapy
Number analyzed (Participants) | 35
Participants | 8

2. Secondary Outcome: Number of Serious Adverse Events.
Description: Assessment of the overall serious adverse event rate.
Time Frame: 2 years
Measure: Number; unit: events
Arm/Group | Intraoperative Radiotherapy
Number analyzed (Participants) | 36
events | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Arm/Group | Intraoperative Radiotherapy
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 6/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Radiotherapy (N=36)
Breast Pain (Reproductive system and breast disorders) | 2
Breast infection/abscess (Skin and subcutaneous tissue disorders) | 1
Edema (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Fibrosis (Skin and subcutaneous tissue disorders) | 1
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Seroma (Musculoskeletal and connective tissue disorders) | 1
Hematoma (Vascular disorders) | 1
urinary retention (Renal and urinary disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-05-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT00556907/Prot_SAP_000.pdf